CLINICAL TRIAL: NCT06246201
Title: An Investigation of The Relationship Between Cognitive Status and Exercise Capacity, Fatigue Perception in Coronary Artery Patients
Brief Title: The Relationship Between Cognitive Status and Exercise Capacity, Fatigue Perception in Coronary Artery Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Saklica, Principal Investigator, Hacettepe University
Other Study IDs: GO 23/639
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
Keywords: Exercise Test; Fatigue; Cognitive Function
MeSH Terms: conditions — Coronary Artery Disease; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Coronary Artery Disease: Having been diagnosed with coronary artery disease

SUMMARY:
The study aimed to examine the relationship between cognitive status, exercise capacity, and fatigue perception in coronary artery disease patients.

DETAILED DESCRIPTION:
Exercise training for patients with coronary artery disease is an essential element of multicomponent cardiac rehabilitation. For the successful implementation of exercise-based cardiac rehabilitation programs, adequate cognitive function (e.g. executive function, selective attention, memory) is an important prerequisite. In patients with atherosclerotic coronary artery disease, the presence of coronary microvascular dysfunction as determined by low coronary flow reserve is associated with abnormal cerebral flow hemodynamics and mild but significant impairment in cognitive function. In the literature, there is no study examining the relationship between cognitive level and fatigue perception.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being diagnosed with coronary artery disease
* To cooperate with the tests to be performed
* Signing a consent form

Exclusion Criteria:

* Presence of neurological disease that may affect cognitive status
* Presence of clinically unstable cardiac disease
* Left ventricular ejection fraction <30%
* Being diagnosed with end-stage renal failure
* Diagnosed with active myocarditis or pericarditis
* Being diagnosed with rhythm disorder
* Having amputation, peripheral arterial disease, musculoskeletal and/or neurological diseases that will prevent participation in functional capacity tests
* Not volunteering to participate in the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are 18 years old and older and are diagnosed with coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Cognitive State Assessment | August 2023-August 2024
  Montreal Cognitive Assessment Scale (MoCA) will be used to assess cognitive status.
Assessment of Exercise Capacity | August 2023-August 2024
  Exercise capacity will be evaluated with modified shuttle walking test.
Assessment of Perceived Fatigue Severity After Exercise Test | August 2023-August 2024
  It will be evaluated on the Modified Borg Scale from 0 to 10. 0 means no fatigue. 10 means extremely tired.

SECONDARY OUTCOMES:
Physical Activity Assessment | August 2023-August 2024
  Physical activity level will be measured with the International Physical Activity Questionnaire (IPAQ). 600 METs (Metabolic Equivalent of Task) min/week means inactive.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Hikmet Yorgun, PhD, Study Chair — Hacettepe University; Ahmet Hakan Ates, PhD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)